CLINICAL TRIAL: NCT02151929
Title: Bioresorbable Vascular Scaffold in Patient With ST Elevation Myocardial Infarction: a Randomized Comparison With Everolimus Eluting Stent
Brief Title: Bioresorbable Vascular Scaffold in Patients With Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Emilio Di Lorenzo MD PhD, Dott. Emilio Di Lorenzo, San Giuseppe Moscati Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM_BVS1
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: ST Elevation Acute Myocardial Infarction
Keywords: myocardial infarction; primary PCI; stent
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable Vascular Scaffold (Experimental): Implantation of of an everolimus eluting bioresorbable scaffold in patients with STEMI treated with primary PCI
  Interventions: Device: Bioresorbable vascular scaffold
- Everolimus Eluting stent (Active Comparator): Implantation of of an everolimus eluting stent in patients with STEMI treated with primary PCI
  Interventions: Device: Everolimus eluting stent

INTERVENTIONS:
Device: Bioresorbable vascular scaffold — stenting of an acute thrombotic lesion in patient within STEMI
  Other Names: BVS, ABSORB (Abbot Vascular)
  Arms: Bioresorbable Vascular Scaffold
Device: Everolimus eluting stent — stenting of an acute thrombotic lesion in patient within STEMI
  Other Names: Xience Prime (Abbott Vascular)
  Arms: Everolimus Eluting stent

SUMMARY:
Evaluation of the feasibility and safety of Bioresorbable Vascular Scaffold (BVS) in patient treated with primary PCI (pPCI).

DETAILED DESCRIPTION:
Background. Drug-eluting stent (DES) implantation may offer benefits in terms of repeat revascularization in patients with ST elevation myocardial infarction (STEMI). The everolimus eluting bioresorbable vascular scaffold (BVS) has shown efficacy and safety in stable patient but not in acute coronary syndromes. The study tested the feasibility and safety of BVS in patient treated with primary PCI (pPCI) Methods. Consecutive STEMI patients admitted within 12 hours of symptom onset and undergoing primary angioplasty and stent implantation at a tertiary center with 24-hour primary PCI capability will be randomly assigned to everolimus eluting stent (EES) or BVS. Primary endpoints are procedural and clinical success. The MACE (cardiac death, non fatal myocardial infarction, target lesion revascularization (TLR)) and definite or probable ST will be evaluated at six months.

ELIGIBILITY:
Inclusion Criteria:

1. chest pain for more than 30 minutes;
2. ST-segment elevation of 1 mm or more in 2 or more contiguous electrocardiograph leads or with presumably new left bundle-branch block

Exclusion Criteria:

1. Active internal bleeding or a history of bleeding diathesis within the previous 30 days;
2. Contraindication to dual antiplatelet therapy for 12 months;
3. Known allergy to everolimus;
4. A history of stroke within 30 days or any history of hemorrhagic stroke;
5. History, symptoms, or findings suggestive of aortic dissection;
6. High-likelihood of death within BVS resorbtion time;
7. Cardiogenic shock;
8. Infarct artery reference diameter, <2.0 mm or >3.7 mm (i.e. not suitable for currently available BVS sizes);
9. Pregnancy;
10. Participation in other trials

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Procedural and Clinical success | Patients will be followed for the duration of hospital stay (4-8 days)
  Procedural success: The deployment of BVS at the intended target lesion with a final residual stenosis ≤20% and a TIMI 2-3 coronary flow by visual estimation without major periprocedural complication (death, emergent CABG, coronary perforation, flow limiting coronary dissection).
  Clinical success: any major in-hospital events (deaths, reinfarction, urgent revascularization, stroke, major bleedings)

SECONDARY OUTCOMES:
The MACE | six months
  cumulative incidence of cardiac death, non fatal myocardial infarction and target lesion revascularization

OTHER OUTCOMES:
stent thrombosis | six months
  cumulative incidence of definite or probable stent thrombosis defined according to the Academic Research Consortium definition

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Di Lorenzo, MD PhD, Principal Investigator — Division of Cardiology AO Moscati Avellino ITALY
Locations (1):
- Division of Cardiology Ao Moscati, Avellino, Italy

REFERENCES:
- [Background] Di Lorenzo E, Carbone G, Sauro L, Casafina A, Capasso M, Sauro R. Bare-metal stents versus drug-eluting stents for primary angioplasty: long-term outcome. Curr Cardiol Rep. 2011 Oct;13(5):459-64. doi: 10.1007/s11886-011-0207-0. PMID 21792636
- [Background] De Luca G, Dirksen MT, Spaulding C, Kelbaek H, Schalij M, Thuesen L, van der Hoeven B, Vink MA, Kaiser C, Musto C, Chechi T, Spaziani G, Diaz de la Llera LS, Pasceri V, Di Lorenzo E, Violini R, Cortese G, Suryapranata H, Stone GW; Drug-Eluting Stent in Primary Angioplasty (DESERT) Cooperation. Drug-eluting vs bare-metal stents in primary angioplasty: a pooled patient-level meta-analysis of randomized trials. Arch Intern Med. 2012 Apr 23;172(8):611-21; discussion 621-2. doi: 10.1001/archinternmed.2012.758. PMID 22529227
- [Background] Di Lorenzo E, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G, De Luca G. Benefits of drug-eluting stents as compared to bare metal stent in ST-segment elevation myocardial infarction: four year results of the PaclitAxel or Sirolimus-Eluting stent vs bare metal stent in primary angiOplasty (PASEO) randomized trial. Am Heart J. 2009 Oct;158(4):e43-50. doi: 10.1016/j.ahj.2009.03.016. PMID 19781402
- [Background] Di Lorenzo E, De Luca G, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G. The PASEO (PaclitAxel or Sirolimus-Eluting Stent Versus Bare Metal Stent in Primary Angioplasty) Randomized Trial. JACC Cardiovasc Interv. 2009 Jun;2(6):515-23. doi: 10.1016/j.jcin.2009.03.012. PMID 19539255
- [Background] Ormiston JA, Serruys PW, Regar E, Dudek D, Thuesen L, Webster MW, Onuma Y, Garcia-Garcia HM, McGreevy R, Veldhof S. A bioabsorbable everolimus-eluting coronary stent system for patients with single de-novo coronary artery lesions (ABSORB): a prospective open-label trial. Lancet. 2008 Mar 15;371(9616):899-907. doi: 10.1016/S0140-6736(08)60415-8. PMID 18342684
- [Background] Serruys PW, Onuma Y, Ormiston JA, de Bruyne B, Regar E, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Miquel-Hebert K, Rapoza R, Garcia-Garcia HM. Evaluation of the second generation of a bioresorbable everolimus drug-eluting vascular scaffold for treatment of de novo coronary artery stenosis: six-month clinical and imaging outcomes. Circulation. 2010 Nov 30;122(22):2301-12. doi: 10.1161/CIRCULATIONAHA.110.970772. Epub 2010 Nov 15. PMID 21098436